CLINICAL TRIAL: NCT06456580
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study With an Open-label Extension Period to Evaluate the Efficacy and Safety of Telitacicept in Patients With Generalized Myasthenia Gravis
Brief Title: A Study of Telitacicept for the Treatment of Generalized Myasthenia Gravis (RemeMG)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vor Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC18G006
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Myasthenia Gravis; gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental): Telitacicept
  Interventions: Biological: Telitacicept
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept — Subcutaneous injection
  Other Names: RC18; RC18-L
  Arms: Telitacicept
Drug: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of telitacicept in the treatment of generalized myasthenia gravis.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is an autoimmune disease that affects the neuromuscular junction on the postsynaptic membrane. The predominant manifestation is muscle weakness, which typically worsens with repeated muscle exertion, such that function is usually the best in the morning with more pronounced weakness at the end of the day. A major challenge in MG is the lack of therapies that cure the disease.

Telitacicept is a fully human TACI-Fc fusion protein that targets B-lymphocyte stimulator (BLyS) and A proliferating-inducing ligand (APRIL), neutralizing their interactions with receptors on B cells. The blockage of BLyS and APRIL interaction with their respective cell membrane receptors (transmembrane activator and CAML interactor [TACI], B-cell maturation antigen, and BLyS receptors) by telitacicept would inhibit B-cell proliferation and maturation. This suppression at the proximal portion of the immune response could alleviate autoimmune symptoms.

This study is a randomized, double-blind, placebo-controlled Phase 3 study with an open-label extension to evaluate the efficacy and safety of telitacicept in a global patient population with gMG.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patient aged ≥18 years at screening.
2. Patients have prior confirmed diagnosis of gMG with generalized muscle weakness (typical pattern of weakness meeting the clinical criteria for diagnosis of MG as defined by the Myasthenia Gravis Foundation of America (MGFA) clinical classification II-IV.
3. Patients have positive antibodies against AChR or MuSK at screening.
4. MG-ADL score ≥6 points at screening and baseline with ocular-related score <50% of the total score.
5. QMG score ≥8 points, and ≥ 4 items score at least 2 points at screening and baseline.

Key Exclusion Criteria:

1. Patients have been diagnosed with any other autoimmune disease which can potentially pose a safety or efficacy confounding risk.
2. Patients having acute or chronic infection.
3. Patients having thymoma within 5 years or received thymectomy ≤6 months prior to screening.
4. Patients having current or history of primary immunodeficiency.
5. Patients having history of malignancy within the last 5 years.
6. Patient having prior or continuing diagnosis of serious cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) score at Week 24 | Week 24
  The MG-ADL is an 8-item patient-reported outcome measure assessing MG symptoms and their effects on daily activities. Each item in the scale is scored on a 0 to 3 (0=normal, 3=severe disease) point scale. The total score is the sum of all individual item scores ranging from 0 to 24. Higher scores indicate more severe disability due to MG. A decrease from Baseline score indicates improvement.

SECONDARY OUTCOMES:
Change from baseline in Quantitative Myasthenia Gravis (QMG) score at Week 24 | Week 24
  The QMG is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The scale consists of 13 items. Each item in the scale is scored on a 0 to 3-point scale, ranging from 0 (no weakness) to 3 (severe weakness), summing up to the overall score range from 0 to 39. Higher scores indicate more severe impairment. A decrease from Baseline score indicates improvement.
Change from baseline in MG Quality of Life scale (MG-QOL15r) at Week 24 | Week 24
  The MG-QoL15r is a 15-item patient-reported outcome measure designed to assess quality of life in patients with MG. Each item in the scale is scored on a 0 to 2-point scale (0=Not at all, 1=Somewhat, 2=Very much). The total score is the sum of the 15 individual item scores, ranging from 0 to 30. Higher scores indicate more severe impact of the disease on aspects of the patient's life. A decrease from Baseline score indicates improvement.
Proportion of patients with a decrease of ≥2 points from baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) score at Week 24 | Week 24
  Proportion of patients with a decrease of ≥2 points from baseline in MG-ADL score at Week 24. The MG-ADL is an 8-item patient-reported outcome measure assessing MG symptoms and their effects on daily activities. Each item in the scale is scored on a 0 to 3 (0=normal, 3=severe disease) point scale. The total score is the sum of all individual item scores ranging from 0 to 24. Higher scores indicate more severe disability due to MG.
Proportion of patients with a decrease of ≥3 points from baseline in Quantitative Myasthenia Gravis (QMG) score at Week 24 | Week 24
  Proportion of patients with a decrease of ≥3 points from baseline in QMG score at Week 24. The QMG is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The scale consists of 13 items. Each item in the scale is scored on a 0 to 3-point scale, ranging from 0 (no weakness) to 3 (severe weakness), summing up to the overall score range from 0 to 39. Higher scores indicate more severe impairment. A decrease from Baseline score indicates improvement.
Proportion of patients who achieved minimal symptomatic expression (MSE, defined as having MG-ADL score of 0 or 1) at Week 24 | Week 24
  Proportion of patients who achieved minimal symptomatic expression (MSE, defined as having MG-ADL score of 0 or 1) at Week 24

CONTACTS AND LOCATIONS:
Locations (84):
- United States (19):
  - University of Southern California, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of California San Francisco (UCSF), San Francisco, California
  - SFM Clinical Research, Boca Raton, Florida
  - Allied Biomedical Research Institute (ABRI), Miami, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Wellstar MCG Health Medical Center, Augusta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville Physicians, Louisville, Kentucky
  - Neurology Center of New England, Foxborough, Massachusetts
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Trinity Health - Grand Rapids Hospital, Grand Rapids, Michigan
  - Mount Sinai Health System, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Health Physicians - Clifton, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - Center for Neurological Disorders, S.C. - Greenfield - Gamma Therapeutic Center, Greenfield, Wisconsin
- Argentina (5):
  - STAT Research S.A., Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital General de Agudos José María Ramos Mejía, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundación Scherbovsky, Mendoza, Mendoza Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Gold Coast University Hospital, Southport, Queensland
- Universitair Ziekenhuis (UZ) Leuven - Campus Gasthuisberg, Leuven, Flemish Brabant, Belgium
- Brazil (5):
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Universidade Estadual de Campinas, Campinas, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Pseg Centro de Pesquisa Clinica, São Paulo, São Paulo
- Canada (2):
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Czechia (3):
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba, Moravian-Silesian
  - MINKSneuro s.r.o. - MUDr. Eduard Minks Ph.D., Brno, South Moravian
  - Fakultni Nemocnice Brno, Brno, South Moravian
- France (2):
  - Hôpital Pasteur, Nice, Alpes-Maritimes
  - Groupe Hospitalier Pellegrin, Bordeaux, Gironde
- Georgia (4):
  - Multi-profile Clinic "New Hospitals", Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
  - Aversi Clinic - Central Branch, Tbilisi
  - Simon Khechinashvili University Hospital, Tbilisi
- Italy (8):
  - IRCCS Fondazione Casa Sollievo della Sofferenza SG Rotondo, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli, Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Napoli
  - Fondazione Istituto San Raffaele - G. Giglio Di Cefalu, Cefalù, Palermo
  - Istituto Neurologico Casimiro Mondino, Pavia, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Rome
  - Azienda Ospedaliera - Universitaria Sant' Andrea, Rome, Rome
- Japan (16):
  - National Hospital Organization - Nagoya Medical Center, Nagoya, Aichi-ken
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Yokohama Medical Center, Yokohama, Kanagawa
  - National Hospital Organization Utano National Hospital, Kyoto, Kyoto
  - NHO Sendai Medical Center, Sendai, Miyagi
  - National Hospital Organization Niigata National Hospital, Kashiwazaki-Shi, Niigata
  - Okinawa National Hospital, Ginowan-Shi, Okinawa
  - Nagoya City University Hospital, Suita-shi, Osaka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Sizuoka [Shizuoka]
  - Tokushima University Hospital, Tokushima, Tokusima [Tokushima]
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
- Poland (11):
  - Niepubliczny Zakład Opieki Zdrowotnej NEURO - KARD, Poznan, Greater Poland Voivodeship
  - Medicover Integrated Clinical Services (MICS) - Centrum Medyczne Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Neurocentrum Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Clinirem - Lublin, Lublin, Lublin Voivodeship
  - Centrum Medyczne Hope Clinic, Lublin, Lubusz Voivodeship
  - Twoja Przychodnia Nowosolskie Centrum Medyczne, Nowa Sól, Lubusz Voivodeship
  - Centrum Medyczne Neuroprot, Warsaw, Masovian Voivodeship
  - MTZ Powered by Pratia, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk, Pomeranian Voivodeship
  - Neurologia Śląska Centrum Medyczne, Katowice, Silesian Voivodeship
- Spain (5):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitari Mútua Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Basurto, Bilbao, Biscay
  - Hospital Universitari i Politècnic La Fe, Valencia, València

IPD SHARING:
Plan to Share IPD: No